CLINICAL TRIAL: NCT06077578
Title: Understanding the Perceptions, Behavior, and Attitudes of Healthcare Professionals, Hospitalized Children, and Parents of These Children Toward Hospital Play Services
Brief Title: Understanding the Perceptions, Behavior, and Attitudes Towards Hospital Play Services
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Li Ho Cheung William, Professor, Chinese University of Hong Kong
Other Study IDs: HPS
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Child Health
Keywords: hospital play services; healthcare professionals; hospitalized children; parents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthcare professionals: Healthcare professionals, including nurses, physicians, physiotherapists, occupational therapists, and radiotherapists, have at least one year experience in caring for hospitalized children will be recruited.
- Previously hospitalized children: Previously hospitalized children who had received a hospital play service provided by hospital play specialists.
- parents: Parents of previously hospitalized children who had received a hospital play service provided by hospital play specialists.

SUMMARY:
Aim This proposed study aims to investigate the perceptions, behavior, and attitudes of healthcare professionals, previously hospitalized children, and parents of these children toward hospital play services in the Hong Kong healthcare system. In addition, in-depth interviews will be conducted with selected participants to investigate their views on the role of hospital play specialists , as well as the sustainability and development of hospital play specialists services in Hong Kong hospitals

Study Design A mixed-methods (quantitative and qualitative) approach will be used to collect data. The study will be divided into two phases. In Phase I, a cross-sectional study, using a structured questionnaire, will be conducted on healthcare professionals in the pediatric units of six acute care public hospitals from different regions of Hong Kong. In Phase II, in-depth semi-structured interviews will be conducted with randomly selected healthcare professionals who have participated in the Phase I study. In addition, the investigators will collect feedback and comments from previously hospitalized children and their parents.

DETAILED DESCRIPTION:
i) Phase I study A retrospective cross-sectional questionnaire will be administered to the healthcare professionals who work in the abovementioned public hospitals. A convenience sample of 182 healthcare professionals will be recruited. In addition, the investigators will contact professional pediatric organizations, such as the Hong Kong Pediatric Society and Hong Kong College of Pediatric Nursing to help invite healthcare professionals to participate in this research.

A structured questionnaire has been developed based on existing international and/or local literature. The information gathered will include perceptions of and attitudes toward hospital play, the feasibility and usefulness of hospital play, understanding the roles and responsibilities of hospital play specialists , perceptions of collaborating with hospital play specialists , and perceptions of the need for hospital play services in Hong Kong hospital settings. In addition, demographic information, including age, gender, occupation, and years of experience in taking care of hospitalized children, will be documented.

Data Analysis for the Phase I Study Data analysis will be performed using SPSS Statistics for Windows, V.26.0 (IBM). Continuous variables with normal distribution will be presented as the mean and standard deviation, and those with non-normal distribution will be presented as the median. Categorical variables will be presented as the frequency and proportion.

ii) Phase II Study A semi-structured interview will be conducted with randomly selected healthcare professionals who have participated in the Phase I study. A semi-structured interview guide will be developed by the research team, which includes a professor with extensive knowledge of and experience in conducting both quantitative and qualitative research related to pediatric patients and hospital play activities and a team of experts working in Playright with extensive experience in conducting hospital play interventions for hospitalized children. The interview guide will be further assessed for its relevancy and wording appropriateness by two advanced practice nurses working in Children's Hospital with extensive experience in providing care for hospitalized children.

A purposive sample of 20 healthcare professionals randomly selected from the Phase I study and 14 children previously admitted to hospitals, and their parents, will be recruited for the interviews. However, the actual sample size will depend on data saturation. A one-to-one audiotaped semi-structured in-depth interview will then be conducted with each participant until data saturation is achieved. Each interview will last approximately 20 to 30 minutes. During each interview, a research assistant will act as the interviewer to facilitate the informants to freely express their feelings, thoughts, and ideas. Another research assistant will act as an observer to document all non-verbal cues of the informants.

Data Analysis for the Phase II Study After conducting the interviews, the recordings will be fully transcribed, verbatim, in Cantonese to capture the nuances of expression unique to the dialect, and selected quotations relevant to the themes will subsequently be translated into English. During the coding process, two researchers will be responsible for analyzing the narratives. The analyses will begin with an intensive examination of the transcripts to search for general constructs and themes. Special attention will be given to constructs that diverge from the major topics framed by the guiding questions. The transcripts will first be coded using the open coding method. Details in the interview conversations will then be closely examined to extract a large number of initial categories. As the number of codes increases, some closely related codes will be merged, resulting in a smaller, more manageable set of codes. Selective coding will then be adopted to code the transcripts using the established categories. To facilitate the data analysis process, meetings will be held to discuss emergent themes. During the coding process, any inconsistencies in the interpretation of quotations or the assignment of codes will be resolved through discussions with the research team members. Finally, a complete set of codes will be generated to facilitate comparisons and the development of themes and categories. To achieve a more coherent and logical structure, the themes and categories will be modified by breaking down complicated concepts, merging similar ones, and rearranging certain themes and categories based on their relationships. The analyses will be performed using NVivo Version 9 (QSR International Pty Ltd., 2010).

To ensure data credibility, the interviewer will first ask iterative questions and use probes during the interviews. Second, debriefing sessions will be held between the research assistants and the principal investigator after every five interviews. Modifications will be made by the principal investigator according to the developing ideas and interpretations. Third, data analysis will be performed by two researchers independently, and field notes will be taken into account during the analysis. Regular research team meetings will be held to resolve any disagreements that may arise. The informants will also be invited to review the transcripts and clarify the meaning of their statements, if required. To increase the transferability of the findings, the study will be conducted in acute care hospitals from different regions in Hong Kong. Purposive sampling will be adopted to maximize sample variation, which will help the investigators to obtain a representative group of informants for the interviews. To ensure the confirmability and dependability of the findings, an audit trail will be maintained by another experienced researcher who is not part of this research team. She will review a collection of documents to attest to the interpretations of the researchers.

ELIGIBILITY:
Healthcare professionals

Inclusion Criteria:

* be aged 18 or above
* be able to read and understand English
* be healthcare professionals, including nurses, physicians, physiotherapists, occupational therapists, and radiotherapists, have at least one year experience in caring for hospitalized children

Exclusion Criteria:

* psychologically or physically unable to communicate

Previously hospitalized children

Inclusion Criteria:

* be aged under 18
* be able to communicate in Cantonese
* be previously hospitalized and had received hospital play service provided by hospital play specialists

Exclusion Criteria:

* psychologically or physically unable to communicate

Parents

Inclusion Criteria:

* be aged 18 or above
* be able to communicate in Cantonese
* his/her children be previously hospitalized and had received hospital play service provided by hospital play specialists

Exclusion Criteria:

* psychologically or physically unable to communicate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 182 healthcare professionals will be recruited in the pediatric units of six acute care public hospitals from different regions of Hong Kong. 14 children previously admitted to hospitals, and their parents, will be recruited in Hong Kong.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Perceptions, behavior, and attitudes | baseline
  The perceptions, behavior, and attitudes of healthcare professionals, previously hospitalized children, and parents of these children toward hospital play services will be investigated by semi-structured in-depth interviews

SECONDARY OUTCOMES:
Perceptions of feasibility and usefulness | baseline
  Perceptions of feasibility and usefulness of healthcare professionals towards hospital play services will be investigated by a structured questionnaire
understanding the roles and responsibilities of hospital play specialists | baseline
  Perceived understanding of healthcare professionals towards the roles and responsibilities of hospital play specialists will be investigated by a structured questionnaire
Perceptions of collaborating with hospital play specialists | baseline
  Perceptions of collaborating with hospital play specialists of healthcare professionals will be be investigated by a structured questionnaire
Perceptions of the need for hospital play services in Hong Kong hospital settings | baseline
  Perceptions of the need for hospital play services in Hong Kong hospital settings of healthcare professionals will be be investigated by a structured questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, Principal Investigator — williamli@cuhk.edu.hk
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The relevant anonymized patient level data, full dataset, technical appendix, and statistical code are available on reasonable request. The approval from the Principal Investigator for the purpose of data use is required.
Time Frame: After the project has been completed and the results of the project has been published
Access Criteria: Request could be sent to Principal Investigator (williamli@cuhk.edu.hk)